CLINICAL TRIAL: NCT03010917
Title: Effect of Fish Oil vs. Placebo on Subjective Effects of Alcohol in Healthy Humans
Brief Title: Fish Oil vs. Placebo on Subjective Effects of Alcohol
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Connecticut Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1609018478
Record Dates: First submitted 2016-12-15; First posted 2017-01-05 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Alcohol Dependence
Keywords: Alcohol Dependence; Fish Oil
MeSH Terms: conditions — Alcoholism | interventions — Fish Oils; Ethanol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fish Oil with ethanol and placebo ethanol infusions (Experimental): Between days 30-40 subjects will participate in 2 test days at least 2 days apart and during the test day will receive an IV infusion of ethanol (placebo vs. targeted Breath Alcohol Concentration ((BrAC) of 100mg%) in a clamped fashion. Test days will be in a randomized order.
  Interventions: Drug: Fish Oil with ethanol and placebo ethanol infusions
- Placebo with ethanol and placebo ethanol infusions (Placebo Comparator): Between days 30-40 subjects will participate in 2 test days at least 2 days apart and during the test day will receive an IV infusion of ethanol (placebo vs. targeted Breath Alcohol Concentration ((BrAC) of 100mg%) in a clamped fashion. Test days will be in a randomized order.
  Interventions: Drug: Placebo with ethanol and placebo ethanol infusions

INTERVENTIONS:
Drug: Fish Oil with ethanol and placebo ethanol infusions — Fish Oil with ethanol and placebo ethanol infusions
  Arms: Fish Oil with ethanol and placebo ethanol infusions
Drug: Placebo with ethanol and placebo ethanol infusions — Placebo with ethanol and placebo ethanol infusions
  Arms: Placebo with ethanol and placebo ethanol infusions

SUMMARY:
This project represents a first step in examining the potential use of fish oil for the treatment of alcohol use disorder (AUD). The investigators will be testing for attenuation of alcohol-induced sedative and stimulant effects, as well as cognitive effects and cerebellar effects in healthy social drinkers.

DETAILED DESCRIPTION:
There have been no studies to date that have examined the relationship between fish oil and alcohol response in humans. The current study was designed to examine the relationship between fish oil and subjective alcohol effects in healthy social drinkers.

This project represents a first step in examining the potential use of fish oil for the treatment of alcohol use disorder (AUD). The investigators will evaluate responses to alcohol through administration of a steady state blood alcohol level (BAL) with an IV infusion using a method that employs an infusion that is titrated to a breathalyzer reading and clamped at a steady state. This approach allows direct comparisons of the acute effects of a specific dose of ethanol between groups, without the confounding factors of variable alcohol absorption and peak BAL's. This approach will allow the examiners to carefully examine if fish oil changes the acute effects of alcohol on a number of outcome domains including subjective drug effects, cognitive performance, and cerebellar effects.

As this study is a pilot study, it is not clear whether fish oil will attenuate alcohol induced subjective stimulation or sedation. Since this is the first study to evaluate fish oil's effects on alcohol-effects in the laboratory, the investigators will be testing for attenuation of alcohol-induced sedative and stimulant effects, as well as cognitive effects and cerebellar effects.

In this study, fish oil will be administered at 3 grams/day for 30-40 days (3 capsules twice a day). The investigators will use 3 grams/day for two reasons: 1) it is within the range of doses safely used in humans (1g to 6g) as a treatment for various psychiatric conditions (depression, anxiety, borderline personality disorder), and 2) is a dose that has shown efficacy in various clinical trials for psychiatric conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females, between the ages of 21 and 55;
2. No current drug use disorder of any drugs of abuse (except tobacco or marijuana);
3. No current medical problems and normal ECG;
4. For women, not pregnant as determined by pregnancy screening nor breast feeding, and using acceptable birth control methods.

Exclusion Criteria:

1. Current major psychiatric illnesses including mood, psychotic, or anxiety disorders;
2. History of major medical illnesses; including liver diseases, heart disease, chronic pain or other medical conditions that the physician investigator deems contraindicated for the subject to be in the study;
3. Liver function tests (ALT or AST) greater than 3 times normal;
4. Allergy to seafood.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-09-08 (Actual)

PRIMARY OUTCOMES:
Assessment of stimulant and sedative effects of alcohol with the Biphasic Alcohol Effects Scale (BAES). | Baseline
  The BAES is a 14-item self-report scale. Seven items measure stimulant effects of alcohol during the test sessions and seven items measure sedative effects. Stimulant and sedative effect scores range from 0 (not at all) to 70 (extremely).
Assessment of stimulant and sedative effects of alcohol with the Biphasic Alcohol Effects Scale (BAES). | Week 4 (test session 1)
Assessment of stimulant and sedative effects of alcohol with the Biphasic Alcohol Effects Scale (BAES). | Week 6 (test session 2)

SECONDARY OUTCOMES:
Cognitive performance measured with the Rapid Information Processing Task (RVIP) | Baseline
  (RVIP) is a widely used task to assess sustained attention, with a working memory component. In this task, a series of single digits is presented on a computer screen at a rate of 100 digits per minute for 4 min. Targets are defined as three consecutive odd digits (e.g., 7-9-3) or three consecutive even digits (e.g., 2-8-6). The percentage of targets correctly detected will be the main outcome measure.
Cognitive performance measured with the Rapid Information Processing Task (RVIP) | Week 4 (test session 1)
  (RVIP) is a widely used task to assess sustained attention, with a working memory component. In this task, a series of single digits is presented on a computer screen at a rate of 100 digits per minute for 4 min. Targets are defined as three consecutive odd digits (e.g., 7-9-3) or three consecutive even digits (e.g., 2-8-6). The percentage of targets correctly detected will be the main outcome measure.
Cognitive performance measured with the Rapid Information Processing Task (RVIP) | Week 6 (test session 2)
  (RVIP) is a widely used task to assess sustained attention, with a working memory component. In this task, a series of single digits is presented on a computer screen at a rate of 100 digits per minute for 4 min. Targets are defined as three consecutive odd digits (e.g., 7-9-3) or three consecutive even digits (e.g., 2-8-6). The percentage of targets correctly detected will be the main outcome measure.
Cognitive performance measured by a "Go No-Go task" will assess the ability to withhold responses to an infrequently occurring target. | Baseline
  A series of blue and green rectangular shapes are presented every 1150 ms and participants are instructed to press a spacebar every time the green rectangular shape appeared, and to give equal importance to speed and accuracy. The primary outcome is the number of errors on the No-Go trials.
Cognitive performance measured by a "Go No-Go task" will assess the ability to withhold responses to an infrequently occurring target. | Week 4 (test session 1)
  A series of blue and green rectangular shapes are presented every 1150 ms and participants are instructed to press a spacebar every time the green rectangular shape appeared, and to give equal importance to speed and accuracy. The primary outcome is the number of errors on the No-Go trials.
Cognitive performance measured by a "Go No-Go task" will assess the ability to withhold responses to an infrequently occurring target. | Week 6 (test session 2)
  A series of blue and green rectangular shapes are presented every 1150 ms and participants are instructed to press a spacebar every time the green rectangular shape appeared, and to give equal importance to speed and accuracy. The primary outcome is the number of errors on the No-Go trials.
Cognitive performance measured by the Hopkins Verbal Learning Test-Revised (HVLT-R). | Baseline
  The HVLT-R is a word list learning test of verbal memory. The outcome is the percent correct on immediate and delayed recall of words on a list.
Cognitive performance measured by the Hopkins Verbal Learning Test-Revised (HVLT-R). | Week 4 (test session 1)
  The HVLT-R is a word list learning test of verbal memory. The outcome is the percent correct on immediate and delayed recall of words on a list.
Cognitive performance measured by the Hopkins Verbal Learning Test-Revised (HVLT-R). | Week 6 (test session 2)
  The HVLT-R is a word list learning test of verbal memory. The outcome is the percent correct on immediate and delayed recall of words on a list.
Motor Impairment: The Grooved Pegboard Test (Lafayette Instrument Company) is a manipulative dexterity test, | Baseline
  This is an eye-to hand timed coordination test. A quicker time indicates greater coordination.
Motor Impairment: The Grooved Pegboard Test (Lafayette Instrument Company) is a manipulative dexterity test, | Week 4 (test session 1)
  This is an eye-to hand timed coordination test. A quicker time indicates greater coordination.
Motor Impairment: The Grooved Pegboard Test (Lafayette Instrument Company) is a manipulative dexterity test, | Week 6 (test session 2)
  This is an eye-to hand timed coordination test. A quicker time indicates greater coordination.

CONTACTS AND LOCATIONS:
Overall Officials: Ismene Petrakis, M.D., Principal Investigator — Yale University/VA Connecticut Healthcare System
Locations (1):
- VA Connecticut Healtcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Subramanian MG, Heil SH, Kruger ML, Collins KL, Buck PO, Zawacki T, Abbey A, Sokol RJ, Diamond MP. A three-stage alcohol clamp procedure in human subjects. Alcohol Clin Exp Res. 2002 Oct;26(10):1479-83. doi: 10.1097/01.ALC.0000034038.41972.36. PMID 12394280
- [Background] Zimmermann US, O'Connor S, Ramchandani VA. Modeling alcohol self-administration in the human laboratory. Curr Top Behav Neurosci. 2013;13:315-53. doi: 10.1007/7854_2011_149. PMID 21792747
- [Background] Ramchandani VA, O'Connor S, Blekher T, Kareken D, Morzorati S, Nurnberger J Jr, Li TK. A preliminary study of acute responses to clamped alcohol concentration and family history of alcoholism. Alcohol Clin Exp Res. 1999 Aug;23(8):1320-30. PMID 10470974